CLINICAL TRIAL: NCT05498259
Title: A Phase 2 Study of Orelabrutinib With R-CHOP-like Regimen for Patients With Newly Diagnosed Untreated Non-GCB DLBCL
Brief Title: Orelabrutinib With R-CHOP-like Regimen for Patients With Newly Diagnosed Untreated Non-GCB DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORIENT
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Orelabrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — orelabrutinib; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib+R-CHOP-like (Experimental): Orelabrutinib plus Rituximab for 21 days; Following Imaging examinations, patients with ≥25% tumor reduction, treat with orelabrutinib 150mg qd orally plus R-CHOP-like for 6 cycles; whereas, patients with <25% tumor reduction, withdraw from the study，treat with R-CHOP-like alone for 6 cycle
  Interventions: Drug: Orelabrutinib; Biological: Rituximab; Drug: CHOP-like Regimen

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib 150mg qd PO
Biological: Rituximab — Rituximab 375 mg/m2 IV on Day 1 of each 21-day cycle
Drug: CHOP-like Regimen — cyclophosphamide, anthracene nucleus chemotherapeutics（doxorubicin，liposomal doxorubicin, etc.）, vinca alkaloids（vincristine, vindesine, etc.），and glucocorticoid （dexamethasone，prednison, etc.）.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of orelabrutinib combined with rituximab，followed by orelabrutinib combined with R-CHOP-like regimen for newly diagnosed untreated Non-GCB DLBCL Patients

DETAILED DESCRIPTION:
The study will start with an initial 21-days of induction therapy with orelabrutinib and rituximab，following imaging examinations to evaluate response rates. Then treatment with 6 cycles chemoimmunotherapy (R-CHOP-like) either alone or in combination with orelabrutinib will depend on response during induction phase. Each cycle is 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Non-GCB DLBCL
2. Age ≥18 and ≤70 years
3. At least one measurable lesion，measurable lymph nodes or masses of at least 15 millimeter (mm)
4. ECOG performance status 0-2
5. Lymphoma International Prognostic Score (IPI) ≥ 2
6. Life expectancy ≥ 6 months
7. Adequate organ and marrow function
8. Agreement to practice birth control from the time of enrollment until the follow-up period of the study

Exclusion Criteria:

1. Received major surgery within 4 weeks before treatment or existed unhealed wounds or ulcers, except biopsy related to lymphoma diagnosis
2. All patients with primary central nervous system lymphoma
3. History of stroke or intracranial hemorrhage within 6 months before screening, require or receive anticoagulant therapy with warfarin or an equivalent antagonist
4. Requires treatment with strong /moderate CYP3A inhibitors or inducers
5. Uncontrolled comorbidity or complications, including but not limited to: symptomatic congestive heart failure (New York Heart Association Class III-IV) or symptomatic or poorly controlled arrhythmias and/or significant pulmonary disease
6. HIV infection and/or active hepatitis B or active hepatitis C infection
7. Uncontrolled active systemic infection
8. Known hypersensitivity or contraindications to any drug involved in the study
9. Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | At the end of Cycle 6（each cycle is 21 days）
  The rate of patients who achieved complete response after treatment by OR-CHOP-like

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | At the end of Cycle 3 and Cycle 6（each cycle is 21 days）
  The rate of patients who achieved CR or PR after treatment by OR-CHOP-like
Progression-free survival（PFS） | up to 24 month after the end of last patient's treatment
  PFS will be assessed from the first OR(Orelabrutinib plus Rituximab) given to date of progression, relapse, death or end of follow-up
Incidence of Treatment-Emergent Adverse Events, Treatment-Related Adverse Events and Serious Adverse Events | initiation of study drug until 30 days after last dose
  The safety and tolerability of the therapeutic regimen measured by the incidence of Treatment-Emergent Adverse Events, Treatment-Related Adverse Events and Serious Adverse Events
Mini response rate | the first 21 days
  The rate of patients who achieve ≥25% tumor reduction after OR treatment

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All the data would be available at the First Affiliated Hospital and other researchers after the end of the study
Supporting Information: Study Protocol, SAP
Time Frame: after the end of the study